CLINICAL TRIAL: NCT04541303
Title: Randomized Study on the Topical Application of Tranexamic Acid to Wound Bed for Hemostasis in the Setting Granulating Wounds Following Mohs Micrographic Surgery
Brief Title: Topical Tranexamic Acid Use on Granulating Wounds Following Mohs Micrographic Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Nicholas J Golda, Principal Investigator, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025444
Record Dates: First submitted 2020-08-28; First posted 2020-09-09 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Wound Haemorrhage
Keywords: tranexamic acid; hemostasis; hemorrhagic complication; bleeding complication; Mohs micrographic surgery; granulating wound; granulating defect
MeSH Terms: interventions — Tranexamic Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: One arm will receive topical application of tranexamic acid (intervention). Other arm with receive topical application of normal saline (placebo).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Physician/surgeon, nurses, patient, and patient family will be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Topical application of tranexamic acid to granulating wound defect status post Mohs micrographic surgery.
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): Topical application of normal saline to granulating wound defect status post Mohs micrographic surgery.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Tranexamic acid — tranexamic acid diluted to concentration of 25ml/mg
  Other Names: Lysteda; Cyclokapron
  Arms: Intervention
Drug: normal saline — 0.9% sodium chloride
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
Bleeding after Mohs micrographic surgery for skin cancer is a low risk complication that can occur. This study aims to determine the effect of a drug, often used to reduce bleeding, called tranexamic acid when applied topically to the skin wound after surgery.

DETAILED DESCRIPTION:
To perform a prospective randomized controlled trial to determine the hemostatic effect of TXA soaked gauze (intervention) versus normal saline soaked gauze (control) when applied to granulating defects in the setting of Mohs micrographic surgery.

Patients meeting inclusion criteria will be randomized into two arms once enrolled in the study on the day of their Mohs micrographic surgery (MMS).

One arm will serve as the control group and will receive normal saline soaked telfa pads to the wound bed upon completion of MMS.

A second arm will receive TXA 25mg/ml at a volume of 1ml/cm2 soaked telfa pads to wound bed upon completion of MMS.

In both arms, the telfa pads will have a standard pressure dressing placed overtop.

ELIGIBILITY:
Inclusion Criteria:

* All adult (18 years or older) patients presenting for Mohs micrographic surgery (MMS) for the treatment of melanoma or nonmelanoma skin cancer (NMSC) with a wound that will be healing by granulation

Exclusion Criteria:

* Patients must not be pregnant or breastfeeding.
* Patients must not have a known allergic reaction or sensitivity to TXA
* Patient must not have an international normalized ratio (INR) out of therapeutic range if on warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Golda, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

REFERENCES:
- [Background] Tolkachjov SN, Brodland DG, Coldiron BM, Fazio MJ, Hruza GJ, Roenigk RK, Rogers HW, Zitelli JA, Winchester DS, Harmon CB. Understanding Mohs Micrographic Surgery: A Review and Practical Guide for the Nondermatologist. Mayo Clin Proc. 2017 Aug;92(8):1261-1271. doi: 10.1016/j.mayocp.2017.04.009. PMID 28778259
- [Background] Kimyai-Asadi A, Goldberg LH, Peterson SR, Silapint S, Jih MH. The incidence of major complications from Mohs micrographic surgery performed in office-based and hospital-based settings. J Am Acad Dermatol. 2005 Oct;53(4):628-34. doi: 10.1016/j.jaad.2005.03.023. PMID 16198783
- [Background] Bunick CG, Aasi SZ. Hemorrhagic complications in dermatologic surgery. Dermatol Ther. 2011 Nov-Dec;24(6):537-50. doi: 10.1111/j.1529-8019.2012.01454.x. PMID 22515669
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Lin ZX, Woolf SK. Safety, Efficacy, and Cost-effectiveness of Tranexamic Acid in Orthopedic Surgery. Orthopedics. 2016 Mar-Apr;39(2):119-30. doi: 10.3928/01477447-20160301-05. Epub 2016 Mar 4. PMID 26942474
- [Background] Roberts I, Shakur H, Coats T, Hunt B, Balogun E, Barnetson L, Cook L, Kawahara T, Perel P, Prieto-Merino D, Ramos M, Cairns J, Guerriero C. The CRASH-2 trial: a randomised controlled trial and economic evaluation of the effects of tranexamic acid on death, vascular occlusive events and transfusion requirement in bleeding trauma patients. Health Technol Assess. 2013 Mar;17(10):1-79. doi: 10.3310/hta17100. PMID 23477634
- [Background] Kagoma YK, Crowther MA, Douketis J, Bhandari M, Eikelboom J, Lim W. Use of antifibrinolytic therapy to reduce transfusion in patients undergoing orthopedic surgery: a systematic review of randomized trials. Thromb Res. 2009 Mar;123(5):687-96. doi: 10.1016/j.thromres.2008.09.015. Epub 2008 Nov 12. PMID 19007970
- [Background] Ausen K, Hagen AI, Ostbyhaug HS, Olafsson S, Kvalsund BJ, Spigset O, Pleym H. Topical moistening of mastectomy wounds with diluted tranexamic acid to reduce bleeding: randomized clinical trial. BJS Open. 2020 Apr;4(2):216-224. doi: 10.1002/bjs5.50248. Epub 2019 Dec 26. PMID 32207575
- [Background] de Vasconcellos SJ, de Santana Santos T, Reinheimer DM, Faria-E-Silva AL, de Melo MF, Martins-Filho PR. Topical application of tranexamic acid in anticoagulated patients undergoing minor oral surgery: A systematic review and meta-analysis of randomized clinical trials. J Craniomaxillofac Surg. 2017 Jan;45(1):20-26. doi: 10.1016/j.jcms.2016.10.001. Epub 2016 Oct 13. PMID 27840121
- [Background] Zahed R, Moharamzadeh P, Alizadeharasi S, Ghasemi A, Saeedi M. A new and rapid method for epistaxis treatment using injectable form of tranexamic acid topically: a randomized controlled trial. Am J Emerg Med. 2013 Sep;31(9):1389-92. doi: 10.1016/j.ajem.2013.06.043. Epub 2013 Jul 30. PMID 23911102
- [Background] Teoh WY, Tan TG, Ng KT, Ong KX, Chan XL, Hung Tsan SE, Wang CY. Prophylactic Topical Tranexamic Acid Versus Placebo in Surgical Patients: A Systematic Review and Meta-analysis *. Ann Surg. 2021 Apr 1;273(4):676-683. doi: 10.1097/SLA.0000000000003896. PMID 32282377
- [Background] Ausen K, Pleym H, Liu J, Hegstad S, Nordgard HB, Pavlovic I, Spigset O. Serum Concentrations and Pharmacokinetics of Tranexamic Acid after Two Means of Topical Administration in Massive Weight Loss Skin-Reducing Surgery. Plast Reconstr Surg. 2019 Jun;143(6):1169e-1178e. doi: 10.1097/PRS.0000000000005620. PMID 31136475
- [Background] Eikebrokk TA, Vassmyr BS, Ausen K, Gravastrand C, Spigset O, Pukstad B. Cytotoxicity and effect on wound re-epithelialization after topical administration of tranexamic acid. BJS Open. 2019 Sep 26;3(6):840-851. doi: 10.1002/bjs5.50192. eCollection 2019 Dec. PMID 31832591
- See also: Ferring Pharmaceuticals Incorporated. Lysteda (tranexamic acid) [package insert]. Revised October 2013. Accessed May 2020. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2013/022430s004lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention - Tranexamic Acid: Topical application of tranexamic acid to granulating wound defect status post Mohs micrographic surgery.
  Tranexamic acid: tranexamic acid diluted to concentration of 25ml/mg
Period: Overall Study
Arm/Group | Intervention - Tranexamic Acid | Placebo
Started | 62 | 62
Completed | 62 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 57 | 56 | 113
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 43 | 47 | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
bleeding [Number; unit: participants] — Patient reported bleeding
  participants | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Postoperative Hemorrhagic Complications
Description: Number of patients who call to report postoperative bleeding
Time Frame: three days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 62 | 62
Participants | 0 | 6
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = .028, None specified

2. Primary Outcome: Rate of Clinic Evaluations of Postoperative Hemorrhagic Complications
Description: The number of patients who return to clinic with postoperative bleeding
Time Frame: three days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Tranexamic Acid | Placebo
Number analyzed (Participants) | 62 | 62
Participants | 0 | 0

3. Primary Outcome: Rate of Treatment Interventions for Postoperative Hemorrhagic Complications
Description: The number of patients who are treated for postoperative bleeding
Time Frame: three days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Tranexamic Acid | Placebo
Number analyzed (Participants) | 62 | 62
Participants | 0 | 1

4. Secondary Outcome: Types of Postoperative Hemorrhagic Complications
Description: postoperative bleeding complications will be defined as arterial bleed, venous oozing, or organized blood clot/hematoma
Time Frame: three days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Tranexamic Acid | Placebo
Number analyzed (Participants) | 62 | 62
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT04541303/Prot_SAP_000.pdf